CLINICAL TRIAL: NCT01692821
Title: Effect of Systemic Hypoxia and Hyperoxia on Retinal Oxygen Saturation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv.-Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OPHT-180312
Record Dates: First submitted 2012-06-14; First posted 2012-09-25 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Retinal Oxygenation; Retinal Blood Flow
Keywords: retinal oxygen saturation; retinal blood flow; hyperoxia; hypoxia
MeSH Terms: conditions — Hyperoxia; Hypoxia | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 100% oxygen breathing (Experimental)
  Interventions: Drug: 100% oxygen breathing
- 15% oxygen in N2 breathing (Experimental)
  Interventions: Drug: 15% oxygen in N2 breathing
- 12% oxygen in N2 breathing (Experimental)
  Interventions: Drug: 12% oxygen in N2 breathing

INTERVENTIONS:
Drug: 100% oxygen breathing — 100% oxygen breathing - 30 minutes
  Arms: 100% oxygen breathing
Drug: 15% oxygen in N2 breathing — 15% oxygen in N2 breathing - 30 minutes
  Arms: 15% oxygen in N2 breathing
Drug: 12% oxygen in N2 breathing — 12% oxygen in N2 breathing - 30 minutes
  Arms: 12% oxygen in N2 breathing

SUMMARY:
Adequate perfusion and oxygenation is essential for the function of the inner retina. Although it is known that oxygen tension is very well autoregulated in the retina, the physiological mechanisms behind this regulation process are not fully explored. The development of new instruments for the non-invasive measurement of oxygen tension in retinal vessels now allows for the more precise investigation of these physiological processes. The current study seeks to evaluate the retinal oxygen saturation in healthy subjects while breathing different oxygen mixtures to achieve a hypoxic and a hyperoxic state.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years
* Nonsmokers
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 3 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study (except oral contraceptive)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence of any form of anemia
* Blood donation during the previous 3 weeks
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Retinal oxygen saturation | On the study day - during each breathing period (6 times)

SECONDARY OUTCOMES:
Retinal blood flow | On the study day - during each breathing period (6 times)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, Assoc. Prof. Priv.-Doz. Dr., Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Palkovits S, Lasta M, Told R, Schmidl D, Boltz A, Napora KJ, Werkmeister RM, Popa-Cherecheanu A, Garhofer G, Schmetterer L. Retinal oxygen metabolism during normoxia and hyperoxia in healthy subjects. Invest Ophthalmol Vis Sci. 2014 Jul 11;55(8):4707-13. doi: 10.1167/iovs.14-14593. PMID 25015353